CLINICAL TRIAL: NCT05780203
Title: The Effects of Exposure in the Context of Anxious Thinking Styles
Brief Title: CBM in the Context of Exposure for Acrophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Beray Macit, PhD Student, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 674
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acrophobia
Keywords: anxiety disorders; acrophobia; exposure; cognitive bias modification; interpretational processing biases
MeSH Terms: conditions — Acrophobia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One session exposure treatment + active Cognitive Bias Modification training (Experimental): The exposure treatment will be administered at the tower of the German Mining museum. The day after the exposure session, patients will complete the CBM training in the lab of the Mental Health and Research Center of Ruhr University Bochum.
  Interventions: Behavioral: One session exposure treatment; Behavioral: Active Cognitive Bias Modification training
- One session exposure treatment + sham Cognitive Bias Modification training (Sham Comparator): The exposure treatment will be administered at the tower of the German Mining museum. The day after the exposure session, patients will complete the sham CBM training in the lab of the Mental Health and Research Center of Ruhr University Bochum.
  Interventions: Behavioral: One session exposure treatment; Behavioral: Sham Cognitive Bias Modification training

INTERVENTIONS:
Behavioral: One session exposure treatment — One session exposure treatment during which patients will be confronted with a height-related situation.
Behavioral: Sham Cognitive Bias Modification training — Sham Cognitive Bias Modification training procedure matched in format to active training but adapted to not target height-related, interpretational processing biases.
  Arms: One session exposure treatment + sham Cognitive Bias Modification training
Behavioral: Active Cognitive Bias Modification training — Active Cognitive Bias Modification training targeting height-related, interpretational processing biases.
  Arms: One session exposure treatment + active Cognitive Bias Modification training

SUMMARY:
The proposed study will apply a one-session exposure treatment combined with CBM training modifying interpretational processing biases versus a sham training in acrophobic individuals. The main aim is to advance our understanding of the mechanisms underlying exposure treatment.

DETAILED DESCRIPTION:
The present study will apply a one-session exposure treatment followed by a computerized interpretational training (CBM) or sham training in acrophobic individuals. By doing so, it aims to better understand the mechanisms underlying exposure, i.e., the role of cognitive change. Specifically, this study aims to enhance changes in disorder-relevant cognitive processing post-exposure, compared to a sham training. Further, we hope to improve both therapy outcomes and the generalization of therapeutic effects.

ELIGIBILITY:
Inclusion criteria:

1. Informed consent
2. Sufficient German language skills to complete the experimental tasks and questionnaires
3. Aged between 18 and 65 years
4. Current primary diagnosis of acrophobia as defined by DSM-5 (based on DIPS)
5. Lives within reasonable travelling distance of the research center

Exclusion criteria:

1. Currently in psychotherapeutic treatment
2. Impaired therapy capability (as judged by researcher/clinician)
3. Current diagnosis of substance use disorder (via DIPS)
4. Current or past diagnosis of psychotic disorder or bipolar disorder (via DIPS)
5. Acute suicidality (via DIPS)
6. Diagnosis of chronical physical or neurological diseases (self-reported by participant)
7. Personality Disorder (via DIPS or via clinical judgement)
8. Attention-deficit hyperactivity disorder (self-reported by participant or via DIPS)
9. Intellectual disability (self-reported by participant or via clinical judgment)
10. Women: pregnancy or breast feeding (self-reported by participant)
11. Intake of medication that could impede the effects of exposure therapy or CBM training (e.g., Lorazepam)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Acrophobia-related interpretational processing biases as measured using the Encoding Recognition Task | baseline, post-training (~1 week post-baseline)
  Acrophobia-related interpretational processing biases will be measured using a modified version of the Encoding Recognition Task (ERT, Salemink & van den Hout, 2010). Bias scores of the Encoding Recognition Task can range from -4 to +4, with lower scores indicating a more negative interpretation bias.
  The primary outcome is change in bias score from baseline to post-training.

SECONDARY OUTCOMES:
Acrophobia-related interpretational processing biases as measured using the Encoding Recognition Task | baseline, pre-training (~1 week post-baseline), follow-up (~5 weeks post-baseline)
  Acrophobia-related interpretational processing biases will be measured using a modified version of the Encoding Recognition Task (ERT, Salemink & van den Hout, 2010). Bias scores of the Encoding Recognition Task can range from -4 to +4, with lower indicating a more negative interpretation bias.
Heights Interpretation Questionnaire (HIQ) | baseline, post-training (~1 week post-baseline), follow-up (~5 weeks post-baseline)
  The Heights Interpretation Questionnaire (HIQ; Steinman & Teachman, 2011) asks participants to rate the likelihood of eight negative interpretations for two height-related, ambiguous scenarios. Scores can range from 16 to 80, with higher scores indicating a worse outcome.
Scrambled Sentences Task (SST) | post-training (~1 week post-baseline), follow-up (~5 weeks post-baseline)
  Modified version of the Scrambled Sentences Task (Wenzlaff & Bates, 1998), including 20 height-related items that can be unscrambled into positive or negative statements.
Danger/ Anxiety Expectancy Scale (DES/AES) | baseline, post-training (~1 week post-baseline), follow-up (~5 weeks post-baseline)
  The Danger/ Anxiety Expectancy Scale (DES/AES; Gursky & Reiss, 1987) asks participants to rate the likelihood of potential harmful events passing through their mind and the likelihood to experience anxiety symptoms if confronted with heights. Scores can range from 15 to 75, with higher scores indicating a worse outcome.
Acrophobia Questionnaire (AQ) | baseline, pre-training (1 day after exposure; ~1 week post-baseline), follow-up (~5 weeks post-baseline)
  The Acrophobia Questionnaire (AQ; Cohen, 1977) asks participants to rate their anxiety and avoidance behavior for 20 common height-related situations. Scores can range from 0 to 160, with higher scores indicating a worse outcome.
Behavioral Approach Task (BAT) | baseline, post-training (~1 week post-baseline), follow-up (~5 weeks post-baseline)
  With the Behavioral Approach Task (BAT), participants' behavioral approach tendencies to height-relevant situations will be assessed by instructing participants to go as high as possible at the emergency staircase at the therapy center and asking participants to rate their subjective fear with the Subjective Units of Distress Scale (SUDS; Wolpe 1973). Scores can range from 0 to 100, with higher scores indicating greater fear.

OTHER OUTCOMES:
Levels of Progesterone and Estradiol | pre-exposure (just before exposure; ~1 week post-baseline)
  Via salivary samples, patients' endogenous levels of estradiol and progesterone will be assessed.
Negative Effects Questionnaire (NEQ) | follow-up (~5 weeks post-baseline)
  Adverse events during the study will be assessed with an adapted version of the Negative Effects Questionnaire, which is a 20-item questionnaire designed to assess potential negative effects of psychological interventions (Rozental et al., 2019), in this context also including the CBM training. Scores can range from 0 to 80, with higher scores indicating more negative effects.
Feedback questionnaire | follow-up (~5 weeks post-baseline)
  We will use a feedback questionnaire containing both rating scales and open questions to assess patients' feedback about the study and interventions completed.
  Scores can range from 21 to 189, with higher scores indicating a more positive feedback.
Depression Anxiety Stress Scale-21 (DASS-21) | baseline
  Symptoms of depression, stress and anxiety will be assessed using the Depression Anxiety Stress Scale-21 (Lovibond & Lovibond, 1995) which consists of seven symptom-related items per subscale. Participants are asked to rate the strength of each symptom in the past week. Scores can range from 0 to 63, with overall higher values indicate more severe symptoms.
High Place Phenomenon Index (HPPI) | baseline
  We will use the High Place Phenomenon Index (HPPI; Hames et al., 2012; German version: Teismann et al., 2020) to assess how often participants experienced the "high place phenomenon". This phenomenon involves the sudden urge to jump down when being in a high place and thus may be relevant in the context of acrophobia. The index consists of three items about three different height-related situations, and patients have to indicate whether they experienced the high place phenomenon in each situation using a 6-point Likert scale. Scores can range from 0 to 15, with higher scores indicating more frequent experiences of the high place phenomenon.

CONTACTS AND LOCATIONS:
Overall Officials: Marcella Woud, Dr., Principal Investigator — marcella.woud@rub.de
Locations (1):
- Mental Health and Research Center, Ruhr University of Bochum, Bochum, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available on publication via a suitable repository such as the Open Science Framework, and will be made available to reviewers at the time of submission (or publically with a pre-print version of the manuscript).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Supporting information will be made available on publication via a suitable repository such as the Open Science Framework, and will be made available to reviewers at the time of submission (or publically with a pre-print version of the manuscript).
Access Criteria: Data made available will be the research data reported in the publication, with the exception of any data that could compromise participant anonymity.
URL: https://osf.io/m35jf/

REFERENCES:
- See also: Project on Open Science Framework — https://osf.io/m35jf/